CLINICAL TRIAL: NCT06857344
Title: Automated Anesthesia System-Gastrointestinal Endoscopy (AAS-GE): a Reinforcement Learning Based Control for Anesthesia During Gastrointestinal Endoscopy
Brief Title: Reinforcement Learned Automatic Anesthesia System During Painless Gastrointestinal Endoscopy
Acronym: AAS-GE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Intelligent Medical Research Center, Shenzhen United Scheme Technology Co., Ltd. (Industry)
Collaborators: Zhengzhou Central Hospital (Other); Xinzheng Public People's Hospital (Unknown); Henan Provincial People's Hospital (Other); Anxi County Hospital (Unknown); Jinjiang Municipal Hospital, Shanghai Sixth People's Hospital Fujian Campus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZUS2025001
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia Induction
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): In the test group, participants will receive anesthesia via an AI model.
  Interventions: Procedure: AI Controlled General Anesthesia
- Control group (Active Comparator): In the control group, anesthesia will be induce by experienced anesthesiologists
  Interventions: Procedure: General Anesthesia (GA)

INTERVENTIONS:
Procedure: AI Controlled General Anesthesia — During gastrointestinal endoscopy, anesthesia will be induced using ciprofol, and controlled by an AI model.
  Arms: Test group
Procedure: General Anesthesia (GA) — Anesthesia will be induced using ciprofol, and controlled by experienced anesthesiologists.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the performance difference between trained model and clinical professionals in anesthesia control during gastrointestinal endoscopy. The participants would include adults aged between 18-65 years old with ASA scores I-II. The main questions it aims to answer are:

* Can AI model successfully and safely perform anesthesia during gastrointestinal endoscopy?
* Researchers hypothesis that anesthesia performed by professionals is not inferior to those performed by AI model.

The researchers will compare the results of the AI group with the traditional group to see if both groups have similar success rates in performing anesthesia.

Participants will fast for 8 hours before the procedure, and drinking water will be prohibited for 2 hours after taking the intestinal purgatives.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class I-II
* Expected operation duration less than 1 hour

Exclusion Criteria:

* History of cardiac, hepatic, renal, or metabolic disorders (e.g., diabetes, hypertension, sleep apnea)
* Known allergy to opioids or ciprofloxacin components
* Cachexia
* Hypothermia; history of narcotic abuse; chronic alcoholism; obesity (BMI >30); patients with apnea
* Current pregnancy or lactation
* History of substance abuse or alcohol dependence
* Participation in any other drug clinical trial within the past 3 months
* Obesity (BMI >30 kg/m²)
* Procedure termination due to gastric retention or inadequate bowel preparation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | During procedure
  Hypoxemia is defined as blood oxygen saturation below 92% at any time.

SECONDARY OUTCOMES:
Area under curve of hypoxemia | During procedure
  The area where SpO2 is below 92%.
Lowest value of blood oxygen saturation | During procedure
Induction and maintenance doses of anesthesia | During procedure
  Doses are recorded in mg/kg/h. The induction period is defined as the interval from the start of anesthesia to the first BIS value below 60. The maintenance period is defined as the interval from the first BIS value below 60 to the end of the drug infusion.
Induction time | During procedure
  The time interval from the start of drug administration to the first BIS ≤ 1.
Complete recovery time | During procedure
  Time interval from cessation of anesthetic agents to BIS > 80.
Incidence of hypotension | During procedure
  systolic blood pressure < 90 mmHg or a 30% decrease from baseline lasting longer than 2 minutes
Counts of body movement | During procedure
Dose of norepinephrine | During procedure
Duration of colonoscopy | During procedure
Ciprofol related adverse reactions | During procedure
  Included sinus bradycardia, dizziness

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anxi County Hospital, Anxi, Fujian
  - Jinjiang Municipal Hospital, Shanghai Sixth People's Hospital Fujian Campus, Jinjiang, Fujian
  - Xinzheng Public People's Hospital, Xinzheng, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided